CLINICAL TRIAL: NCT03861247
Title: Individualized Treatment of Hyperphosphatemia Based on Phosphate Balance in Maintenance Hemodialysis Patients: a Multicenter, Randomized Clinical Trial
Brief Title: Individualized Treatment of Hyperphosphatemia in Maintenance Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chen Jing (Other)
Collaborators: Huadong Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Chen Jing, Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2018470
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Maintenance Hemodialysis; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Drug: Phosphate-binder intervention
- Intervention group (Experimental)
  Interventions: Drug: Phosphate-binder intervention; Dietary Supplement: Phosphorus-restricted dietary intervention

INTERVENTIONS:
Drug: Phosphate-binder intervention — Use phosphate-binders according to KDIGO Guidelines, Chinese Guidance for Diagnosis and Treatment of Mineral and Bone Disorder in Chronic Kidney Disease and drug specification .
Dietary Supplement: Phosphorus-restricted dietary intervention — Use low phosphorus diet and prolong the time of hemodialysis according to the phosphorus balance evaluation if necessary
  Other Names: Additional dialysis intervention
  Arms: Intervention group

SUMMARY:
The research is designed as a prospective, randomized, controlled clinical trial without blinding. A total of 116 participants with hyperphosphatemia will be enrolled from three hemodialysis center (56 from Huashan Hospital, 30 from Huadong Hospital and 30 from Tongji Hospital). All participants will be randomly divided into control group and intervention group in a ratio of 1:1. Phosphorus balance status is evaluated in participants of the intervention group by the phosphorus balance calculator. Then, these participants will be given individualized phosphate-binders, dietary and dialysis intervention according to the results of phosphorus balance evaluation. Participants in the control group will not receive the phosphorus balance status evaluation but receive phosphate-binder treatment according to the KDIGO Guidelines. Dietary phosphorus intake, dialysate calcium concentration and dose of active vitamin D, phosphorus-binders of all participants will be recorded during the whole research program. After two-week treatment, the phosphorus balance of participants in intervention group will be evaluated again and the therapeutic strategies then will be adjusted. At the same time, the therapeutic strategies of participants in the control group will be adjusted according to the serum phosphorus concentration. All participants will be followed up for two weeks again and receive blood test and related examinations at the end of study. The results of final examinations will be analyzed to evaluate the efficacy of individualized treatment of hyperphosphatemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject within 18-85 years old, male or female.
2. Subject receiving maintenance hemodialysis 3 times weekly at least 3 months with autologous arteriovenous fistula.
3. Subject with hyperphosphatemia as defined by serum phosphorus concentration >1.45mmol/L.
4. Subject in a good general condition with a stable dietary habit.
5. Subject has insight of the disease and treatment himself/herself and haves ability to communicate with others.
6. Subject has provided informed consent.

Exclusion Criteria:

1. Subject has residual renal function.
2. Subject with severe infection, anemia (Hb<60g/L) or hypoproteinemia (Alb<30g/L).
3. Subject has cancer or cachexia.
4. Subject with a history of myocardial infarction, coronary angioplasty, or coronary arterial bypass grafting within the past 3 months.
5. Subject with severe hematopoietic system disease, such as aplastic anemia, thalassemia and thrombocytopenic purpura.
6. Subject with severe gastrointestinal system disease such as dysphagia, hypohepatia, Active gastrointestinal bleeding, ileus, enterobrosis, or received subtotal gastrectomy.
7. Subject with disease which affects serum phosphorus concentration such as hypoparathyroidism (iPTH<11pg/ml), severe hyperparathyroidism (iPTH>600pg/ml) and type 2 vitamin D dependence rickets.
8. Subject is pregnant.
9. Subject is currently enrolled in or has completed any other investigational device or drug study<30 days prior to screening, or is receiving other investigational agents.
10. Subject has inadequate hemodialysis with a recent spKt/V<1.2.
11. Subject has a poor nutritional status with a recent (nPNA<1.0g/kg/d) .
12. Subject is not a good participant for the research in the opinion of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus concentration | Four weeks after treatment
Achievement rate of serum phosphorus | Four weeks after treatment

SECONDARY OUTCOMES:
Serum calcium concentration | Four weeks after treatment
Serum iPTH concentration | Four weeks after treatment
Serum albumin concentration | Four weeks after treatment

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huadong Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital, Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No